CLINICAL TRIAL: NCT05397548
Title: Use of Circulating Exosomal lncRNA-GC1 as Blood Biomarker for Early Detection and Monitoring Gastric Cancer
Brief Title: Use of Circulating Exosomal LncRNA-GC1 to Monitor Gastric Cancer
Acronym: UCELMGC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lin Chen (Other)
Collaborators: Xijing Hospital (Other)
Responsible Party: Sponsor-Investigator, Lin Chen, Vice Director of Department of General Surgery, Chinese PLA General Hospital, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: GC-biomarker
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Gastric Cancer
Keywords: Circulating exosomal lncRNA-GC1; Advanced Gastric Carcinoma; early detection; progression
MeSH Terms: conditions — Stomach Neoplasms; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: Gastric cancer cases from two medical centers in China
  Interventions: Diagnostic Test: Measurement of levels of circulating exosomal lncRNA-GC1
- control: Controls from two medical centers in China
  Interventions: Diagnostic Test: Measurement of levels of circulating exosomal lncRNA-GC1

INTERVENTIONS:
Diagnostic Test: Measurement of levels of circulating exosomal lncRNA-GC1 — Each participant was enrolled to assess the levels of circulating exosomal lncRNA-GC1

SUMMARY:
Background:

Although its incidence and mortality has decreased, gastric cancer (GC) is the fourth most common cancer and the second leading cause of cancer-related death worldwide, particularly in China. The number of new cases and deaths may comprise approximately one-half of the global total. The high mortality of GC is partially attributed to late detection and nonspecific symptoms. The current gold standard for diagnosing GC is endoscopic biopsy. However, because of its discomfort to the patient and high cost, screening for early GC (EGC) is a major difficulty in clinical practice, particularly for asymptomatic individuals. Unfortunately, gastric precursor lesions such as intestinal metaplasia (IM), chronic atrophic gastritis (CAG), and persistent Helicobacter pylori (HP) infection increase the difficulty of screening for EGC. Furthermore, the standard serum biomarkers for GC, such as CEA, CA72-4, and CA19-9 achieve a low positive rate. Thus, it is critically important to develop new approaches for diagnosing EGC with high specificity and sensitivity.

Objective:

To study circulating exosomal lncRNA-GC1 as a potential biomarker for detection of gastric cancer.

Eligibility:

Participants from two medical centers in China

Design:

Investigators will use blood samples from participants in the two medical centers. Investigators will use samples from some who developed gastric cancer. The other samples will be from some who stayed cancer free in that time.

Participants already gave written informed consent.

Investigators will take exosomes from the samples and look for lncRNA-GC1.

DETAILED DESCRIPTION:
Late detection is a major reason for the poor prognosis of patients with gastric cancer. For example, the proportion of patients diagnosed with early gastric cancer is as low as 9% in China. The survival rate of patients with early gastric cancer ranges from 60%-80% compared with 15%-24% of patients with advanced gastric cancer. It is therefore imperative to develop novel, relatively noninvasive approaches to improve early diagnosis of gastric cancer. Endoscopy has been considered as the gold standard for diagnosis of gastric cancer but endoscopy-based mass screening may not be feasible in relatively low-risk or less developed regions. Therefore, identification of biomarkers for early stage disease is crucial to in the development of effective screening strategies. With the recent advances in cancer genetics and assay technologies, this is an opportune time to discover minimally invasive, specific, and cost-effective biomarkers. The investigators' previous study has identified circulating exosomal lncRNA-GC1 as a potential biomarker for gastric cancer. The investigators then conducted this prospective study to further investigate the predictive value of circulating exosomal lncRNA-GC1 for early-detection and monitoring progression of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* Histologically confirmed gastric adenocarcinoma

Exclusion Criteria:

* Other previous malignancy within 5 year
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study
* Pregnancy or lactation period
* Legal incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample Shanxi - Hospital and community sample Beijing -Hospital
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Detection of levels of circulating exosomal lncRNA-GC1 | Through study completion, an average of 1 year
  Levels of circulating exosomal lncRNA-GC1 are detected by RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Qiying Song, MD, Study Director — Chinese PLA General Hospital
Locations (1):
- Xinxin Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared until the final results published.